CLINICAL TRIAL: NCT05011630
Title: Specific Bile Microorganisms Caused Intra-abdominal Abscess on Pancreaticoduodenectomy Patients: Customized Antibiotics And Antifungal Medication May Be Necessary
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201803035RIND
Record Dates: First submitted 2021-08-15; First posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Intraabdominal Abscess After Procedure
Keywords: pancreaticoduodenectomy, biliary drainage, positive bile culture, intra-abdominal abscess, surgical complication
MeSH Terms: conditions — Abdominal Abscess | interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IAA group: Intraabdominal abscess (IAA) is defined as either a turbid discharge from the intraoperatively placed drain or a postoperative fluid collection managed by CT-guided placement of drains with documental bacteriological culture.
  Interventions: Other: Pancreaticoduodenectomy
- Non-IAA group: No IAA formation
  Interventions: Other: Pancreaticoduodenectomy

INTERVENTIONS:
Other: Pancreaticoduodenectomy — The incidece of IAA after pancreaticoduodectomy; to validate the risk factors of IAA

SUMMARY:
Background Intra-abdominal abscess (IAA) is one of the most serious surgical infectious complications on pancreaticoduodenectomy (PD) patients. Preoperative biliary drainage (PBD) is considered as a risk of surgical infectious complications. However, the reason why PBD caused IAA was unknown. In this study, we hypothesize that bile contamination may increase the rate of IAA as bile from residual common bile duct (CBD) leaks and contaminates the abdominal cavity.

Methods We retrospectively collected PD patients with performance of bile culture between 2007 and 2019 in our institute. As to bile culture, we used a swab to do intraoperative bile cultures after transection of the CBD. IAA was defined as a postoperative fluid collection managed by CT-guided placement of drains with documental bacteriological culture.

ELIGIBILITY:
Inclusion Criteria:

* all pancreaticoduodenectomy patients

Exclusion Criteria:

* no bile cultures

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical populations
Sampling Method: Non-Probability Sample
Enrollment: 539 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Intraabdominal abscess | 1 month after surgery
  The abscess formation after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Ming Wu, MD, Principal Investigator — National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: No